CLINICAL TRIAL: NCT06562725
Title: Ventilator Settings for Bronchoscopy During Mechanical Ventilation: a Randomized Controlled Study
Acronym: VentSetFib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-01
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation Complication; Fiberoptic Bronchoscopy; Critical Illness; Acute Respiratory Failure
Keywords: Fiberoptic bronchoscopy; Mechanical Ventilation; acute respiratory failure; Tracheostomy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard ventilator settings (No Intervention): Patients randomized in the control group "standard ventilator settings" will be left on the ventilator settings previously chosen by the attending physician, except Inspired Oxygen Fraction(FiO2) increased to 100%
- specific ventilator settings (Experimental): Patients randomized in the experimental group "special ventilator settings" will receive ventilator settings aimed at reducing airway pressure during FOB. This includes : inspiratory flow <25 L/min, tidal volume = 5 mL/Kg, inspiratory time = 1 sec, respiratory frequency <20c/min, PEEP = 5 cmH2O, and FiO2 = 100%
  Interventions: Other: specific ventilator settings

INTERVENTIONS:
Other: specific ventilator settings — The special ventilator settings used in the intervention group - aimed at reducing airway pressure - include inspiratory flow <25 L/min, tidal volume = 5m L/Kg, inspiratory time = 1 sec, respiratory frequency <20 c/min, PEEP = 5 cmH2O, and FiO2 = 100%
  Arms: specific ventilator settings

SUMMARY:
Fiberoptic bronchoscopy (FOB) can cause a significant increase in respiratory resistances and airway pressure during mechanical ventilation (MV), which can jeopardize the delivery of the ventilatory assistance. This randomized controlled study tests the hypothesis that new ventilator settings aimed at reducing airway pressure may facilitate FOB during MV. Results of this trial should lead to propose a new ventilatory strategy for critically ill patients needing a FOB procedure under MV.

DETAILED DESCRIPTION:
Introduction : Fiberoptic bronchoscopy (FOB) during mechanical ventilation (MV) is a challenging procedure as it considerably reduces the endotracheal tube internal diameter, increasing respiratory resistances, which may compromise the delivering of the ventilatory assistance. According to respiratory physiology principles applied to MV, the reduction of inspiratory flow and tidal volume are likely to reduce airway pressure during the inspiratory phase when respiratory resistances increase. Based on this assumption, we propose new ventilator settings aimed at reducing airway pressure during FOB. This study represents the first investigation to test special ventilator settings in order to facilitate FOB during MV.

Methods and analysis : This is a single-center randomized controlled trial, in which intubated patients undergoing a FOB will be assigned (1/1) either to receive the new ventilatory strategy or to stay on the ventilator settings previously selected by the attending physician. The intervention group will be applied the specific ventilator settings (inspiratory flow <25 L/min, tidal volume = 5 mL/Kg, inspiratory time = 1 sec, respiratory frequency <20c/min, positive end expiratory pressure(PEEP) = 5 cmH2O). The primary endpoint will be the reduction of the occurrence of a serious adverse event - inability to deliver the ventilatory support, significant arterial desaturation, or hemodynamics instability - during FOB prompting the interruption of the procedure. The sample size was estimated at a minimum of 46 patients to demonstrate a 50% reduction in the occurrence of such a serious adverse event with a power of 90% and an alpha risk of 0.05 (paired Student t-test).

An adjudication committee evaluates images (scope and monitor) to validate primary endpoint. This is done blinding randomization group.

Results of this trial should lead to propose a new ventilatory strategy for critically ill patients needing a FOB procedure under MV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Acute respiratory failure requiring invasive mechanical ventilation in the intensive care unit;
* Indication of either a fiberoptic bronchoscopy (FOB) procedure or a percutaneous tracheostomy under FOB control;
* Patient under sedation with Richmond Agitation and Sedation Scale(RASS) ≤-2,
* Written informed consent obtained by the patient or the patient legal representative

Exclusion Criteria:

* Presence of an absolute contraindication to FOB (respiratory arrest, severe acute respiratory distress syndrome (ARDS), refractory shock, uncontrolled heart rhythm disorder);
* Patients in respiratory distress or with severe patient-ventilator desynchronies ;
* Patients refusing FOB;
* Pregnancy ;
* Moribund patients (according to American Society of Anesthesiologists (ASA) Physical status score classification, class 5: high probability of death within 24 hours) or at high risk of death during the FOB procedure;
* Patients deprived of liberty;
* Patients under curators or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Determine if the use of specific ventilator settings facilitates the performance of fiberoptic bronchoscopy (FOB) during mechanical ventilation compared to conventional ventilator settings. | 5 minutes after bronchoscopy initiation
  Occurrence of a serious adverse - ventilatory, respiratory, or circulatory - event prompting the procedure to be interrupted early in the first 5 minutes.

SECONDARY OUTCOMES:
determine if the specific ventilator settings prevent significant hypoventilation during FOB | 5 minutes after bronchoscopy initiation
  Significant reduction in minute ventilation during FOB compared to its initial value
determine if the specific ventilator settings prevent significant arterial oxygen desaturation during FOB | 5 minutes after bronchoscopy initiation
  Significant decrease in the "partial pressure of oxygen in arterial blood (PaO2)"/FiO2 ratio during FOB compared to its initial value
determine if the specific ventilator settings prevent significant hypercapnia during FOB | 5 minutes after bronchoscopy initiation
  Significant increase in PaCO2 during FOB compared to its initial value
determine if the specific ventilator settings reduce the incidence of hemodynamic adverse event | 5 minutes after bronchoscopy initiation
  Significant reduction in episodes of tachycardia, arrythmia, or circulatory instability occurring during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm LEMYZE, Dr, Principal Investigator — arras hospital
Locations (1):
- Arras Hospital, Arras, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemyze M, Granier M, Laouki CE, Belmeguenai A, Chared H, Audegond C, Mallat J. Ventilator settings for fibreoptic bronchoscopy during mechanical ventilation: a study protocol for a pragmatic randomised double-blind controlled trial VentSetFib. BMJ Open. 2025 Feb 26;15(2):e096164. doi: 10.1136/bmjopen-2024-096164. PMID 40010841